CLINICAL TRIAL: NCT03208465
Title: Empagliflozin Versus Sitagliptin Therapy for Improvement of Myocardial Perfusion Reserve in Diabetic Patients With Coronary Artery disease_ELITE Trial
Brief Title: Empagliflozin Versus Sitagliptin Therapy for Improvement of Myocardial Perfusion Reserve in Diabetic Patients With Coronary Artery Disease
Acronym: ELITE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: CHEOL WHAN LEE, M.D., Ph.D (Other)
Responsible Party: Sponsor-Investigator, CHEOL WHAN LEE, M.D., Ph.D, professor, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMCCV2016-20
Record Dates: First submitted 2017-06-28; First posted 2017-07-05 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Diabetes Mellitus; Coronary Disease
Keywords: Empagliflozin; Sitagliptin; Myocardial perfusion reserve
MeSH Terms: conditions — Diabetes Mellitus; Coronary Disease | interventions — empagliflozin; Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with Empagliflozin (Experimental)
  Interventions: Drug: Empagliflozin
- Patients with Sitagliptin (Active Comparator)
  Interventions: Drug: Sitagliptin

INTERVENTIONS:
Drug: Empagliflozin — In empagliflozin group, patients will be prescribed empagliflozin 10mg/day.
  Arms: Patients with Empagliflozin
Drug: Sitagliptin — In sitagliptin group, patients will be prescribed sitagliptin 100mg/day.
  Arms: Patients with Sitagliptin

SUMMARY:
This trial evaluates the effects of Empagliflozin versus Sitagliptin, in addition to standard of care, on global myocardial perfusion reserve using dynamic single-photon emission computed tomography (SPECT) images.

ELIGIBILITY:
Inclusion Criteria:

* Men or women at least 19 years of age
* Type 2 diabetes mellitus
* Stable coronary artery disease
* Global myocardial perfusion reserve (MPR) index < 2.5
* The patient or guardian agrees to the study protocol and the schedule of clinical and dynamic SPECT follow-up, and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethical Committee of the respective clinical site.

Exclusion Criteria:

* Contraindications to empagliflozin, Sitagliptin
* DPP4 inhibitors or Sodium-glucose cotransporter-2(SGLT2) inhibitors within the previous 4 weeks
* Insulin requiring diabetes
* Poor glucose control (HbA1C>10 %)
* Acute coronary syndrome
* Stent placement within the previous 6 months
* Previous coronary artery bypass graft surgery within the previous 6 months
* Planned revascularization within 6 months
* Heart failure requiring loop diuretics
* Severe left ventricular hypertrophy (left ventricular septal wall thickness > 13mm)
* Significant renal disease manifested by creatinine clearance of < 30 ml/min)
* Hepatic disease or biliary tract obstruction, or significant hepatic enzyme elevation (alanine transaminase or Aspartate Aminotransferase > 3 times upper limit of normal)
* Radiopaque material implanted in the chest wall (metal, silicone, etc.)
* Contraindication to adenosine stress test
* Any clinically significant abnormality identified at the screening visit, physical examination, laboratory tests, or electrocardiogram which, in the judgment of the Investigator, would preclude safe completion of the study.
* Patient's pregnant or breast-feeding or child-bearing potential
* Expected life expectancy < 1 year
* Unwillingness or inability to comply with the procedures described in this protocol

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-08-07 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Percent change in global myocardial perfusion reserve (MPR) index | 6 months
  Percent change in global myocardial perfusion reserve (MPR) index defined as (global MPR index at 6 months - global MPR index at baseline)/(global MPR index at baseline)x100.
  MPR index=stress myocardial flow/rest myocardial flow

SECONDARY OUTCOMES:
Percent change in regional MPR index | 6 months
  Percent change in regional MPR index defined as (regional MPR index at 6 months - regional MPR index at baseline)/(regional MPR index at baseline)x100.
Absolute change in regional MPR index | 6 months
Absolute change in global MPR index | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Oh M, Choi JH, Kim SO, Lee PH, Ahn JM, Lee SW, Moon DH, Lee CW. Comparison of empagliflozin and sitagliptin therapy on myocardial perfusion reserve in diabetic patients with coronary artery disease. Nucl Med Commun. 2021 Sep 1;42(9):972-978. doi: 10.1097/MNM.0000000000001429. PMID 34397987